CLINICAL TRIAL: NCT05749471
Title: Sexual Dysfunction in Patients With Chronic Venous Disease
Brief Title: Sex Dysfunction and Chronic Venous Disease
Acronym: SEXVENO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2018.61
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Chronic Venous Insufficiency; Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic venous disease: Consecutive patients with chronic venous disease (CVD) that will be diagnosed, staged according to the CEAP (Clinical-Etiology-Anatomy-Pathophysiology) classification of CVD. ASEX (Arizona Sexual Experience) questionnaire will be administered to CVD patients at time 0 of study inclusion and after treatment of CVD at intervals of 6 months and 12 months after treatment.
  Interventions: Diagnostic Test: ASEX (Arizona Sexual Experience) administration

INTERVENTIONS:
Diagnostic Test: ASEX (Arizona Sexual Experience) administration — ASEX is a five-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Possible total scores range from 5 to 30. Generally, a subject with a total ASEX score of > 19, any one item with a score of > 5, or any three items with a score of > 4 would have sexual dysfunction.

SUMMARY:
Chronic Venous Disease (CVD) is a common clinical condition with a high prevalence in the western population that may affect quality of life (QoL) of affected patients for several adverse effects. Sexual dysfunction (SD) also partecipate in the QoL of people and has never specifically studied in CVD patients. The aim of this study is to study SD in CVD patients before and after treatment.

DETAILED DESCRIPTION:
Chronic Venous Disease (CVD) is a widespread clinical condition with a high prevalence in the western world, affecting more than 10% in young adults and more than 70% in older individuals (age >70 years). CVD clinical manifestations vary from mild clinical signs, including varicose veins, to more advanced and severe signs such as. Lower limb edema, skin changes, and venous leg ulceration (VLU) which impact the quality of life (QoL) of affected patients. Sexual dysfunction (SD), generally affects QoL, and specifically SD has never been evaluated in CVD patients. Clinical stages are described by the CEAP (Clinical-Etiology-Anatomy-Pathophysiology) classification that is an internationally accepted standard for describing patients with CVD. CEAP defines the following clinical classes, C0 includes no visible or palpable signs of venous disease; C1 includes telangiectasia and reticular veins; C2 includes trunk VV of variable origin; C2r includes recurrent varicose veins; C3 includes lower limbs edema; C4a includes pigmentation or eczema; C4b includes lipodermatosclerosis or atrophie blanche; C4c includes corona phlebectatica; C5 includes healed ulcer; C6 includes active ulcer; C6r includes recurrent active ulcer. Moreover, each clinical class may be subcharacterized by a subscript indicating the presence (symptomatic, s) or absence (asymptomatic, a) of symptoms attributable to venous disease, such as leg heaviness, achy or tired legs, cramping, restless legs. The most severe form of CVD is defined Chronic Venous Insufficiency (CVI) and corresponds to C3-C6 classes of CEAP. For the treatment of CVD several strategy, often combined can be used such as the administration of vasoactive drugs (VADs), or the utilization of compression devices (elastic stockings or bandages) and several surgical or endovascular techniques.

Regarding sex dysfunction there are several unidimensional self-report measures available for assessing sexual dysfunction, all of them with some advantages and limitations. One of the most scale used in this context, proved useful in several clinical contexts is the ASEX (Arizona Sexual Experience) scale that is considered extremely reliable, valid, and sensitive for measuring sexual dysfunction with optimal internal consistency. ASEX is a five-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Possible total scores range from 5 to 30. Generally, a subject with a total ASEX score of > 19, any one item with a score of > 5, or any three items with a score of > 4 would have sexual dysfunction.

The aim of this study is to evaluate sexual functioning with ASEX scale among patients with CVD, at various clinical stages, before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

- patients with first diagnosis of Chronic Venous Disease

Exclusion Criteria:

* presence of known sexual dysfunction of organic origin.
* presence of arterial system diseases.
* presence of malignancies.
* presence of endocrine system disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sex, with minimum age of 18, with first diagnosis of Chronic Venous Disease.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sexual dysfunction at CVD diagnosis | 6 months
  CVD patients will be evaluated for sexual dysfunction at the moment of first diagnosis of CVD. ASEX (Arizona Sexual Experience) scale will be used. ASEX is a five-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Possible total scores range from 5 to 30. Generally, a subject with a total ASEX score of > 19, any one item with a score of > 5, or any three items with a score of > 4 would have sexual dysfunction

SECONDARY OUTCOMES:
Evolution od sexual dysfunction after CVD treatments | 12 months
  CVD patients that resulted affected from sexual dysfunction related to CVD conditions, will be evaluated to find out if CVD treatment has been beneficial also to sexual dysfunction. ASEX (Arizona Sexual Experience) scale will be used as in outcome 1.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D.; P.h.D., Principal Investigator — University Magna Graecia of Catanzaro
Locations (1):
- University Magna Graecia of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elnazer HY, Baldwin DS. Structured review of the use of the Arizona sexual experiences scale in clinical settings. Hum Psychopharmacol. 2020 May;35(3):e2730. doi: 10.1002/hup.2730. Epub 2020 Mar 31. PMID 32236977
- [Result] Costa D, Andreucci M, Ielapi N, Serraino GF, Mastroroberto P, Bracale UM, Serra R. Molecular Determinants of Chronic Venous Disease: A Comprehensive Review. Int J Mol Sci. 2023 Jan 18;24(3):1928. doi: 10.3390/ijms24031928. PMID 36768250
- [Result] Agaba PA, Ocheke AN, Akanbi MO, Gimba ZM, Ukeagbu J, Mallum BD, Agaba EI. Sexual Functioning and Health-related Quality of Life in Men. Niger Med J. 2017 May-Jun;58(3):96-100. doi: 10.4103/nmj.NMJ_225_16. PMID 29962650
- [Result] Boyacioglu NE, Oflaz F, Karaahmet AY, Hodaei BK, Afsin Y, Tasabat SE. Sexuality, quality of life and psychological well-being in older adults: A correlational study. Eur J Obstet Gynecol Reprod Biol X. 2023 Jan 12;17:100177. doi: 10.1016/j.eurox.2023.100177. eCollection 2023 Mar. PMID 36718173
- [Result] McGahuey CA, Gelenberg AJ, Laukes CA, Moreno FA, Delgado PL, McKnight KM, Manber R. The Arizona Sexual Experience Scale (ASEX): reliability and validity. J Sex Marital Ther. 2000 Jan-Mar;26(1):25-40. doi: 10.1080/009262300278623. PMID 10693114